CLINICAL TRIAL: NCT05966402
Title: Evaluation of Immersion in Virtual Reality in the Management of Anxiety, Then Pain, of Patients in Interventional Imaging.
Acronym: IRVARI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 19-197
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Interventional Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental)
  Interventions: Other: Virtual Reality
- standard care (No Intervention)

INTERVENTIONS:
Other: Virtual Reality — Immersion in Virtual Reality
  Arms: Virtual Reality

SUMMARY:
Investigators propose to use static VR scenarios, adapted to the patient's preferences (sea, mountain, countryside…) to immerse them in an emotionally positive environment. The objective is to reduce the anxiety and pain associated with IR acts in the operating room.

Hypothesis tested:

The use of the 3D immersion of an oculus rift DK2 virtual reality headset during an interventional radiology intervention would reduce the anxiety felt by patients by 25%, evaluated by the STAI YB scale. The correlation between the STAI YB and the APAIS and HAD scales will also be tested.

ELIGIBILITY:
Inclusion Criteria:

* Patients (18-80 years old) with an indication for performing one of the following interventional radiology procedures, according to HAS recommendations: Liver biopsy puncture, embolization of varicoceles, embolization of pelvic varices, embolization of uterine fibroids, Hepatic arterial chemoembolization for hepatocellular carcinoma, radioembolization.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Minor or age > 80 years.
* People suffering from psychiatric pathologies, chronic depressive syndrome or chronic anxiety disorder.
* People with a high risk of motion sickness during virtual reality immersion (MMSQ and VIMSSQ > 80th percentile).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
anxiety measured with STAI Y-B | once (as close as possible to the interventional gesture, i.e. just after it.)
  For the main objective, the STAI Y-B will be used to assess reactive anxiety as close as possible to the interventional gesture, i.e. just after it.

CONTACTS AND LOCATIONS:
Locations (1):
- CAEN University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No